CLINICAL TRIAL: NCT07138235
Title: Complications of Laparoscopic Hiatal Hernia Repair Complicated by Gastroesophageal Reflux Disease Using the ERAS Protocol
Acronym: hiatal hernia
Status: Completed | Type: Observational
Sponsor: Osh State University (Other)
Collaborators: Kyrgyz State Medical Academy (Other)
Responsible Party: Principal Investigator, Zhypargul Abdullaeva, PhD, Lecturer, Osh State University
Other Study IDs: Laparoscopic hiatal hernia
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hiatal Hernia; Hiatal Hernia With Gastroesophageal Reflux Disease
Keywords: laparoscopic hiatal hernia repair,; ERAS protocol,; surgical outcomes
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Procedure: laparoscopic hiatal hernia repair — Intraoperative endoscopic control and the use of calibration bougies allow for increasing the accuracy of cardiac sphincter reconstruction and reducing the risk of hyper- or hypocorrection. Endoscopic equipment. The Olympus EVIS EXERA III endoscopic video system (Olympus Medical Systems Corp., Tokyo, Japan), series 190, was used for diagnostic and therapeutic endoscopic examinations.
  The complex included:
  * CV-190 video processor with digital image magnification,
  * CLV-190 light source (xenon/LED), providing high brightness and uniformity of illumination, a high definition (HD) video monitor,
  * GIF-HQ190, GIF-H190 high-resolution series gastroscopes,
  * CF-HQ190L/I series colonoscopes (if necessary). These functions made it possible to more accurately assess the condition of the mucous membrane of the esophagus and stomach, as well as to identify pathological changes.
  Medications: omeprazole/esomeprazole, ondansetron, cephalosporins intravenously, metoclopramide.

SUMMARY:
Nissen fundoplication with cruroraphy performed according to ERAS protocols in patients with HH complicated by GERD.

DETAILED DESCRIPTION:
The surgery was performed in accordance with the following stages. Preparation for surgery included premedication, thromboembolic prophylaxis, and intravenous administration of broad-spectrum antibiotics 30 minutes before induction of anesthesia. Patient position and approaches: the patient was on the operating table in the spinal position with the lower limbs abducted, the head was raised by 15-20° to improve visualization of the subdiaphragmatic space. Four ports were used: one 10-mm port in the umbilical region (for optics), two 5 mm ports in the right hypochondrium and epigastrium, and one 10 mm port in the left hypochondrium. Based on the analysis of early experience of laparoscopic interventions in the cardioesophageal zone, we modified the standard port technique. In particular, the rejection of the classic fan-shaped installation of five trocars turned out to be justified, since two trocars in the left hypochondrium anatomically conflict and limit the maneuverability of the instruments, also the use of an ultrasonic dissector, allowing for simultaneous coagulation and dissection of tissue, which significantly reduced the need for an additional assistant instrument. This ensured more ergonomic manipulations, reduced the duration of the operation and the need for an additional fifth port.

ELIGIBILITY:
Inclusion Criteria: were clinically significant hiatal hernia complicated by GERD, confirmed endoscopically and by radiological methods, age from 18 to 80 years and ineffectiveness of drug therapy for more than 6 months.

-

Exclusion Criteria: were patients who had previously undergone surgery on the upper abdominal organs and oncological diseases. All patients underwent a comprehensive preoperative examination, including general clinical and biochemical tests, ECG, endoscopy and X-ray of the esophagus, stomach and duodenum.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 106 patients with grade III-IV HH complicated by GERD, who underwent laparoscopic cruroraphy and Nissen fundoplication using the ERAS protocol.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
decreased complication rate and high patient satisfaction | October 2016 to June 2025

IPD SHARING:
Plan to Share IPD: No